CLINICAL TRIAL: NCT06671028
Title: Ropivacaine Versus Ropivacaine with Lidocaine Mixture in Poplitial-Sciatic Nerve Block for Below Knee Surgeries- a Randomized, Single Center Study
Brief Title: Mixed Local for Sciatic Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Cheng Lin, Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 125572
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Regional Anesthesia; Local Anesthetic
MeSH Terms: interventions — Ropivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Active Comparator): Popliteal block using Ropivacaine 100 mg in 20 mL
  Interventions: Drug: Ropivacaine 0,5%
- Ropivacaine anmd Lidocaine (Experimental): Popliteal sciatic block using Ropivacaine 100 mg and Lidocaine 100 mg in 20 mL
  Interventions: Drug: Ropivacaine and Lidocaine

INTERVENTIONS:
Drug: Ropivacaine and Lidocaine — Popliteal sciatic block using Ropivacaine 100 mg and Lidocaine 100 mg in 20 mL
  Arms: Ropivacaine anmd Lidocaine
Drug: Ropivacaine 0,5% — Popliteal sciatic block using ropivacaine 0.5% 20 mL
  Arms: Ropivacaine

SUMMARY:
Choice of local anesthetics is the major determinant of the characteristics of a peripheral nerve block. Short acting local anesthetics while provides faster onset suffer from shorter duration. On the other hand, long acting local anesthetics while provides long duration suffered from long onset time. The ideal local anesthetics should provide faster nerve block onset while providing reasonable duration to provide sustained postoperative analgesia. Mixing short and long acting local anesthetics for nerve blocks may appear to be the solution however previous published studies have demonstrated similar onset time to long acting local anesthetics and with reduced duration. Recently, the London Health Sciences Centre established an ambulatory surgical centre. Fast onset peripheral nerve block is desirable. Previous studies have not looked at popliteal sciatic block and anecdotally we feel addition of short acting local anesthetics appear to speed up onset. We are therefore interested in conducting a randomize trial to determine whether mixing short and long acting local anesthetics can speed up onset of surgical quality block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Scheduled for elective below-knee surgeries such as ankle arthroscopy, lower limb fracture fixation, toe surgeries, etc
* Capable of providing informed consent

Exclusion Criteria:

* History of allergic reaction to local anesthetics
* Pre-existing neurological disorders affecting lower limbs
* Significant renal or hepatic impairment
* Pregnancy or breastfeeding
* Less than 60kg
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete sensory block | Tested every 2 min up to 60 min
  The primary outcome is onset time for achievement of complete sensory block of the sciatic nerve determined via pinch test.

SECONDARY OUTCOMES:
Duration of analgesia | up to 48 hours after discharge
  Patient self reported time to onset of pain or analgesics
Pain score at 6 hour post-block | 6 hours after nerve block
  Numeric rating scale of patient self-reported pain at 6 hour after block placement
Patient satisfaction | at 48 hour
  5 point categorical

IPD SHARING:
Plan to Share IPD: Undecided
This will require REb approval

REFERENCES:
- [Background] Bugamelli S, Zangheri E, Montebugnoli M, Borghi B, Ricci A, De Simone N, Bonfatti M, Elmar K, Luppi M, Pignotti E. One-day surgery for acquired forefoot deformity: sciatic nerve blockade with mepivacaine vs mepivacaine+ropivacaine: a prospective, randomized study. Minerva Anestesiol. 2007 Jan-Feb;73(1-2):57-64. PMID 17356507
- [Background] Cuvillon P, Nouvellon E, Ripart J, Boyer JC, Dehour L, Mahamat A, L'hermite J, Boisson C, Vialles N, Lefrant JY, de La Coussaye JE. A comparison of the pharmacodynamics and pharmacokinetics of bupivacaine, ropivacaine (with epinephrine) and their equal volume mixtures with lidocaine used for femoral and sciatic nerve blocks: a double-blind randomized study. Anesth Analg. 2009 Feb;108(2):641-9. doi: 10.1213/ane.0b013e31819237f8. PMID 19151302
- [Background] Valery P, Aliaksei M. A comparison of the onset time of complete blockade of the sciatic nerve in the application of ropivacaine and its equal volumes mixture with lidocaine: a double-blind randomized study. Korean J Anesthesiol. 2013 Jul;65(1):42-7. doi: 10.4097/kjae.2013.65.1.42. Epub 2013 Jul 19. PMID 23904938
- [Background] Chen L, Wang Q, Shi K, Liu F, Liu L, Ni J, Fang X, Xu X. The effects of lidocaine used in sciatic nerve on the pharmacodynamics and pharmacokinetics of ropivacaine in sciatic nerve combined with lumbar plexus blockade: a double-blind, randomized study. Basic Clin Pharmacol Toxicol. 2013 Mar;112(3):203-8. doi: 10.1111/bcpt.12008. Epub 2012 Dec 6. PMID 22985391